CLINICAL TRIAL: NCT00943904
Title: Comparison of Motor and Sensory Response With Interstim Stimulation for Overactive Bladder and Urgency-Frequency Syndrome
Brief Title: Comparison of Motor and Sensory Response With Interstim Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Karen Noblett, Division Director, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-6799
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-08

CONDITIONS: Overactive Bladder; Urgency-Frequency
Keywords: urinary leakage associated with urinary urgency; unable to fully empty bladder; Comparison: Motor&Sensory Response to Interstim Stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interstim stimulation (Experimental): Patients who receive the interstim implant in order to evaluate effectiveness of treatment
  Interventions: Device: Interstim implant for SNS

INTERVENTIONS:
Device: Interstim implant for SNS — stimulates third sacral nerve root
  Other Names: Sacral nerve Stimulation

SUMMARY:
Sacral nerve stimulation (SNS) implantation is a minimally invasive procedure which has current FDA approval for urinary urge incontinence, urgency-frequency syndrome and non-obstructive urinary retention, and has been available in the United States since 1997. The SNS delivers non-painful, mild electrical pulses to the sacral nerves to modulate the reflexes that influence the bladder, sphincter, and pelvic floor to improve or restore normal voiding function. While SNS has been shown to have efficacy for the aforementioned conditions, the exact mechanism of action is unknown, but it is believed to work primarily through the somatic afferent system in promoting inhibitory reflex pathways to facilitate urine storage. The degree of stimulation is thought to be at a level that only evokes a sensory and not a motor response; however this has not been tested.

DETAILED DESCRIPTION:
SNS involves a two-stage procedure. The initial phase is considered the test stimulation period where the patient is allowed to evaluate whether or not the therapy is effective in controlling her symptoms. There are two techniques that exist in performing the test stimulation. The first is an office-based procedure termed the percutaneous nerve evaluation (PNE). This involves placing a temporary electrode wire through the S3 sacral foramen under local anesthesia. The wire is secured with tape and connected to an external generator the patient wears for a trial period of 3-7 days. If patients have at least 50% improvement in their symptoms during the test phase, they are candidates for chronic implant of the lead and implantable pulse generator (IPG). The advantage of the PNE is that it is an incision free procedure performed in the office utilizing local anesthesia, and does not require hospitalization. The disadvantage comes from the fact that the wire is not securely anchored in place, and has the propensity to migrate away from the nerve with physical activity. The second alternative is known as a staged implant. This is typically performed as an outpatient procedure using local anesthesia, intravenous sedation, and intra-operative fluoroscopy. This procedure involves placement of the chronic quadripolar lead wire adjacent to a sacral nerve root (typically S3). The lead is self-anchoring and therefore reduces the potential for migration. The patient goes through a test phase that can last from 7-21 days. The advantage of this technique is that it allows for a longer trial period with minimal risk of lead migration. The chronic wire also has 4 electrodes that can each be trialed as the active electrode to achieve optimal improvement in patients' symptoms. In addition, during the 2nd stage, or final implant the previously placed tined-lead remains in place and is simply connected to the IPG. This eliminates the chance of variable lead placement from the test and implantation phases. The disadvantage of the staged implant is that it requires two visits to the operating room and may be more costly to the health care system. However, in a prospective study comparing the PNE to the staged implant, there was a significantly higher rate of conversion to implant with the staged procedure vs. the PNE (88% vs.46%). In addition, infection rates are not higher with the staged implant when compared to the PNE.

ELIGIBILITY:
Inclusion Criteria:

* You are eligible to participate in this study if:

  * you are at least 18 years of age or older
  * you have the capacity to give informed consent
  * you are currently implanted with a functioning Interstim device for the treatment of urge urinary leakage or overactive bladder

Exclusion Criteria:

* You are not eligible to participate in this study if:

  * you do not meet the inclusion criteria and/or are not able to fully empty your bladder
  * you have a history of an underlying neurologic disorder
  * you are currently pregnant, or have an active urinary tract or vaginal infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Women's Healthcare, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interstim Stimulation
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interstim Stimulation
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Percent of Symptoms With Improvement of Leaks Reported
Description: Percent change in improvement of symptoms after reprogramming in terms of number of leaks reported. Nocturia refers to leaks that happened while asleep. Incontinence refers to both stress and urge leaks. Urgency refers to only urge leaks. Positive values represent more improvement of symptoms and therefore less leaks. Negative values represent less improvement and therefore more leaks.
Time Frame: 6 months following enrollment
Measure: Number; unit: Percent change in leaks
Arm/Group | Interstim Stimulation
Number analyzed (Participants) | 31
Percent change in leaks
  Nocturia | 14.4
  Incontinence | 19.8
  Urgency | 18.2

ADVERSE EVENTS:
Arm/Group | Interstim Stimulation
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No